CLINICAL TRIAL: NCT00163475
Title: The MOVE-study: Morning Versus Evening Administration of 500 mcg Roflumilast Once Daily for 6 Weeks in Patients With Asthma
Brief Title: Efficacy and Safety of Roflumilast Taken in the Morning or Evening in Patients With Stable Asthma (12 to 70 y) (BY217/M2-015)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-015
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Asthma; Roflumilast
MeSH Terms: conditions — Asthma | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
Bronchial asthma is among the world's most prevalent diseases. Roflumilast is a novel, orally active, selective enzyme inhibitor (phosphodiesterase 4 inhibitor), which has shown effectiveness in the treatment of asthma.

The aim of the study is to compare the effect of roflumilast on lung function, symptoms, and use of rescue medication in patients with stable asthma. Roflumilast will be administered orally either in the morning or in the evening at one dose level. The study duration consists of a baseline period (1 to 2 weeks) and a treatment period (6 weeks). The study will provide further data on safety, tolerability, and effectiveness of roflumilast.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Diagnosis of persistent bronchial asthma (with reference to the Global Initiative for Asthma Guidelines 2002)
* Baseline FEV1 50 - 85% in patients either untreated or receiving e.g. short-acting bronchodilators, DSCG, nedocromil, anticholinergics, long-acting bronchodilators, theophylline/aminophylline, lipoxygenase inhibitors, leukotriene antagonists, alone or in combination
* Baseline FEV1 60 - 90% in patients receiving not more than 500 mcg BDP-CFC (or equivalent) and/or in combination with any other asthma medication mentioned above
* No change in the asthma treatment 4 weeks prior to baseline period
* Patients who, with the exception of asthma, are in good health

Main Exclusion Criteria:

* Poorly controlled asthma: requirement of a course of oral and/or parenteral glucocorticosteroids 4 weeks prior to the baseline, or admission to hospital for asthma (including treatment in an emergency room) 4 weeks prior to the baseline period, or asthma exacerbation in the last 4 weeks prior to baseline period
* Patient using regularly >8 puffs/day rescue medication prior to baseline
* History of lower airway infection in the last 4 weeks prior to baseline period
* Diagnosis of chronic obstructive pulmonary disease and/or other relevant lung diseases
* Heavy smoker: currently: >20 cigarettes/day and/or >10 pack years, ex-smoker: with a smoking history of ≥10 pack years
* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation
* Liver insufficiency (Child Pugh A or worse)
* Active hepatitis
* Known infection with HIV
* Diagnosis or history of cancer (other than basal cell carcinoma) or recurrence within 5 years prior to study start
* Alcohol and/or drug abuse
* Suspected hypersensitivity and/or contraindication to any ingredients of the study medication (roflumilast) or rescue medication
* Pregnancy or patient of childbearing potential who is not using reliable method of contraception
* Patients not able to follow study procedures, e.g. due to language problems, psychological disorders
* Suspected inability or unwillingness to comply with the study procedures

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 511
Dates: Start 2004-05; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
mean change from randomization to endpoint in forced expiratory volume in one second.

SECONDARY OUTCOMES:
forced expiratory vital capacity
peak expiratory flow
morning and evening peak expiratory flow (patient's diary)
symptom score and use of rescue medication (patient's diary)
Asthma Control Questionnaire (ACQ)
proportion of symptom-free days / rescue medication-free days asthma exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (5):
- ALTANA Pharma, Cities in Australia, Australia
- ALTANA Pharma, Cities in Belgium, Belgium
- ALTANA Pharma, Cities in France, France
- ALTANA Pharma, Cities in South Africa, South Africa
- ALTANA Pharma, Cities in Spain, Spain

REFERENCES:
- [Derived] Bateman ED, Bousquet J, Aubier M, Bredenbroker D, O'Byrne PM. Roflumilast for asthma: Efficacy findings in non-placebo-controlled comparator and dosing studies. Pulm Pharmacol Ther. 2015 Dec;35 Suppl:S11-9. doi: 10.1016/j.pupt.2015.10.002. Epub 2015 Oct 8. PMID 26456372
- See also: BY217-M2-015-RDS-2006-06-09 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4473&filename=BY217-M2-015-RDS-2006-06-09.pdf